CLINICAL TRIAL: NCT02377063
Title: Study of the Effect of Fruit/Vegetable Based Supplementation on Microbiome
Brief Title: The Effect of Fruit/Vegetable Drinks on the Human Intestine
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Zhaoping Li, Professor of Medicine, University of California, Los Angeles
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 15-000274
Record Dates: First submitted 2015-02-18; First posted 2015-03-03 (Estimated); Results first posted 2019-09-09 (Actual); Last update posted 2019-09-09 (Actual); Status verified 2019-08

CONDITIONS: Intestinal Bacteria Flora Disturbance
Keywords: colonic flora; microbiomes
MeSH Terms: interventions — Fruit

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- pressed juice 6 bottles (Other): Subjects will consume pressed juice daily for 3 days.
  Interventions: Dietary Supplement: Pressed Juice

INTERVENTIONS:
Dietary Supplement: Pressed Juice — Subjects will be taking vegetable/fruit juice supplementation for 3 days. Blood, urine and stool samples will be collected at baseline, day 4 and day 17.
  Other Names: Fruit/vegetable supplement

SUMMARY:
This is a 4 ½ week study with 20 healthy subjects (including a 2 week run-in ) . Subjects will be taking vegetable/fruit juice supplementation for 3 days. Blood, urine and stool samples will be collected at baseline, day 4 and day 17. The purpose of the study is to determine the effects of fruit/vegetable supplementation on colonic flora.

DETAILED DESCRIPTION:
A total of 20 subjects will be recruited from The UCLA Center for Human Nutrition/Clinical Trials Unit database, print and/or radio advertisements, UCLA campus wide e-mail, the clinicaltrials.gov website, and flyers posted on campus and in the community.

Interested persons will call a telephone number dedicated to the study where they will be instructed to leave their name and phone number. These individuals will be contacted by a study staff member, who will briefly describe the study and answer any questions to ascertain interest. If the individual is interested they will be asked to complete a brief pre-screen form over the telephone to establish eligibility. Individuals who remain interested will be invited for a screening visit. Pre-screen surveys for those not eligible will be shredded.

At screening, informed consent and HIPAA authorization will be reviewed and signed prior to any procedures being done, a medical history will be obtained. If subjects are healthy by medical history the following procedures will be conducted:

* a fasting blood sample will be collected for routine safety labs (CBC and Chemistry Panel)
* complete medical and medication history
* brief physical examination (including vital signs, height and weight)
* Dietary instruction to limit consumption of <3 servings of fruit and vegetables, vitamins and antibiotics
* Dispense materials to collect fecal sample

Results will be reviewed by the study physician for compliance to inclusion and exclusion criteria and the subject will be collected and instructed whether or not they are eligible and should proceed with the stool collection after 2 weeks of dietary compliance. Once the collection is obtained subjects will be asked to return to the clinic in 24 hours.

Baseline, days 4 and 17

During the study visits, the following assessments will be conducted:

* Vital signs, body weight
* Collect fecal sample
* Fasting blood sample
* 24 hour urine
* Dispense materials to collect fecal sample
* Dispense study supplement (Baseline and Day 17 only)
* Assess for compliance of study supplement
* Instructions on symptom diary
* General well-being questionnaire
* Subjects who are compliant will be given a 3-day supply of fruit/vegetable juice at the end of the study

Subjects will be instructed to start with their first juice upon waking or when the normally eat breakfast at intervals of approximately two hours throughout the day. Five (5) 16oz. juices and one (1) 16oz almond milk drink will be numbered and subjects will be asked to consume the product in the numbered sequence. Subjects will be instructed to avoid alcohol, caffeine, and nicotine and hydrate by drinking 8 glasses of water per day for the duration of the study. If needed, subjects will be allowed to drink a cup of herbal tea, water with lemon, almonds, cucumber or an apple during the fruit/juice supplementation.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-50 years of age at screen
2. Subjects must read and sign the Institutional Review Board-approved written informed consent prior to the initiation of any study specific procedures or enrollment. A subject will be excluded for any condition that might compromise the ability to give truly informed consent.

Exclusion Criteria:

1. Any subject with a history of diabetes mellitus on medications, hyperlipidemia on medications, or other serious medical condition, such as chronic hepatic or renal disease, bleeding disorder, congestive heart disease, chronic diarrhea disorders, myocardial infarction, coronary artery bypass graft, angioplasty within 6 months prior to screening, current diagnosis of uncontrolled hypertension (defined as systolic BP>160mmHg, diastolic BP>95mmHg), active or chronic gastrointestinal disorders, bulimia, anorexia, or endocrine diseases (except thyroid disease requiring medication) as indicated by medical history or routine physical examination.
2. Any subject with a screening laboratory value outside of the laboratory normal range that is considered clinically significant for study participation by the investigator.
3. Any subject who currently uses tobacco products.
4. Any history of gastrointestinal disease except for appendectomy
5. No antibiotics or laxatives use during the 2 months before the study.
6. Any allergies to nuts
7. Any subject who is unable or unwilling to comply with the study protocol.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2015-04; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Zhaoping Li, M.D., Ph.D., Principal Investigator — UCLA Department of Medicine, Division of Clinical Nutrition
Locations (1):
- UCLA Center for Human Nutrition, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: UCLA IRB-approved flyers were posted around campus. Interested subjects who respond to the approved flyers called the research site and a coordinator conducted a screening by utilizing the screening script. Eligible subjects will be scheduled for a screening visit began 5/12/2015- 7/7/2015.
Groups:
- Pressed Juice: Subjects will consume pressed juice supplementation for 3 days
  Pressed Juice: Subjects will be taking vegetable/fruit juice supplementation for 3 days. Blood, urine and stool samples will be collected at baseline, day 4 and day 17.
Period: Overall Study
Arm/Group | Pressed Juice
Started | 25
Completed | 20
Not Completed | 5
Not completed — Non-compliance | 5

BASELINE CHARACTERISTICS:
Arm/Group | Pressed Juice
Number analyzed (Participants) | 25
Age, Categorical [Count of Participants; unit: Participants] — Population: Five subjects who did not provide fecal samples were excluded from the analysis.
  Participants
    <=18 years | 0
    Between 18 and 65 years | 25
    >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19
  Male | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 11
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 10
  More than one race | 2
  Unknown or Not Reported | 1

OUTCOME MEASURES:

1. Primary Outcome: Change in Colonic Flora Composition
Description: Changes in microbial count (%) were calculated as the values at day 4 minus the values at baseline
Time Frame: baseline and day 4
Population: All participants for whom colonic flora composition were measured at baseline and day 4.
Measure: Mean (Standard Error); unit: percentage of total bacteria
Groups:
- Mixed Fruit and Vegetable Juice 6 Bottles: All participants consumed 6 bottles of mixed fruit and vegetable juice daily for 3 days.
Arm/Group | Mixed Fruit and Vegetable Juice 6 Bottles
Number analyzed (Participants) | 20
percentage of total bacteria
  Phylum Firmicutes at day 0 | 52.4 (3.9)
  Phylum Firmicutes at day 4 | 41.2 (3.5)
  Phylum Bacteroidetes at day 0 | 41.4 (3.8)
  Phylum Bacteroidetes at day 4 | 51.9 (3.5)
Statistical Analysis 1: Comparison: Mixed Fruit and Vegetable Juice 6 Bottles; Comparison was made to day 4 minus day 0 (baseline) change of phylum Firmicutes after juice consumption; Test type: Other; p = 0.014, ANOVA — p<0.05 was defined as significant; Mean Difference (Final Values) = -11.2
Statistical Analysis 2: Comparison: Mixed Fruit and Vegetable Juice 6 Bottles; Comparison was made to day 4 minus day 0 (baseline) change of phylum Bacteroidetes after juice consumption; Test type: Other; p = 0.026, ANOVA — p<0.05 was defined as significant; Mean Difference (Final Values) = 10.5

ADVERSE EVENTS:
Time Frame: 17 days
Arm/Group | Pressed Juice
All-Cause Mortality (participants affected / at risk) | 0/25
Serious Adverse Events (participants affected / at risk) | 0/25
Other Adverse Events (participants affected / at risk) | 0/25

LIMITATIONS AND CAVEATS:
The study did not address the mechanistic aspect of juice-induced colonic flora composition change.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes